CLINICAL TRIAL: NCT07352982
Title: Effect of Transcutaneous Tibial Nerve Stimulation on Women With Primary Dysmenorrhea
Brief Title: Transcutaneous Tibial Nerve Stimulation on Women With Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Amira Rashad Mohamed Darwish, B.Sc. in Physical Therapy, Pharos University in Alexandria, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-685
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Transcutaneous Tibial Nerve Stimulation; Women; Primary Dysmenorrhea
MeSH Terms: interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (group A) (Experimental): Patients will receive the transcutaneous tibial nerve stimulation (TTNS) and traditional treatment (Nonsteroidal anti-inflammatory drugs) for three sessions a week for four consecutive weeks.
  Interventions: Other: Transcutaneous tibial nerve stimulation (TTNS)
- Control group (group B) (Active Comparator): Patients will receive the placebo transcutaneous tibial nerve stimulation (TTNS) and traditional treatment (Nonsteroidal anti-inflammatory drugs) for three sessions a week for four consecutive weeks.
  Interventions: Drug: Traditional treatment (Nonsteroidal anti-inflammatory drugs)

INTERVENTIONS:
Other: Transcutaneous tibial nerve stimulation (TTNS) — Patients will receive the transcutaneous tibial nerve stimulation (TTNS) and traditional treatment (Nonsteroidal anti-inflammatory drugs) for three sessions a week for four consecutive weeks.
  Arms: Study group (group A)
Drug: Traditional treatment (Nonsteroidal anti-inflammatory drugs) — Patients will receive the placebo transcutaneous tibial nerve stimulation (TTNS) and traditional treatment (Nonsteroidal anti-inflammatory drugs) for three sessions a week for four consecutive weeks.
  Arms: Control group (group B)

SUMMARY:
This study aims to investigate the effects of transcutaneous tibial nerve stimulation (TTNS) on women with primary dysmenorrhea (PD).

DETAILED DESCRIPTION:
Dysmenorrhea is defined as painful menstrual cramps of uterine origin, and considered as one of the most common gynecological disorders among females of childbearing age.

Primary dysmenorrhea (PD) typically manifests within 6-12 months following menarche. It is not associated with organic lesions but is primarily attributed to uterine smooth muscle spasms and vasoconstriction, which are induced by elevated prostaglandin levels.

Additionally, the use of transcutaneous tibial nerve stimulation (TTNS), which consists of the stimulation of the posterior tibial nerve in the superomedial region of the ankle, may be a promising treatment option. The hypogastric sympathetic plexus (L4-L5) and the pelvic parasympathetic plexus (S2-S4) have the same medullar level as the posterior tibial nerve (L4-S3). Thus, inhibitory and excitatory impulses that control the function of the pelvic viscera at the level of the spinal cord can be rebalanced with their stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 20-25 years old.
* Body mass index (BMI) doesn't exceed 30 kg/m2.
* Patients referred from a Gynecologist with a diagnosis of Primary Dysmenorrhea (PD).
* Patients have regular menstrual cycles.
* Patients suffer from pain located in the suprapubic area, abdomen, lower lumbar area, perineum, and/or medial aspect of the thighs during at least half of their annual menstrual cycles and/or in the last 3 cycles.

Exclusion Criteria:

* Patients diagnosed with gynecological pathology.
* Patients taking oral contraceptives or had an intrauterine device implanted.
* Patients had bad obstetric situations or diseases that could interfere with participation.
* Patients have certain disorders including uncorrected coagulopathies, severe comorbid disorder, cancer in the last 5 years or at present, presence of erosions on the inner aspect of the ankle, severe mental disorders, or neuropathies affecting the lower limb.
* Patients who are smoking or taking oral sedatives.
* Patients had undergone surgery or childbirth in the last 6 months.
* Patients who are pregnant.

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women With Primary Dysmenorrhea
Enrollment: 32 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 6 months after the procedure
  Pain Intensity will be assessed using visual Analogue Scale (VAS). VAS consisted of a continuous 10 cm line that represents the pain intensity, ranging from zero; on the left side, which indicates no pain, or discomfort to 10; on the right side, which indicates the worst possible pain he could feel.

SECONDARY OUTCOMES:
Prostaglandin level | 6 months after the procedure
  Serum Prostaglandin will be measured.
Assessment of Quality of Life | 6 months after the procedure
  Quality of Life (QOL) will be assessed using the Arabic Version of the Short Form 36 Health Questionnaire. This questionnaire will be used for assessment of QOL. It is made up of 35 items that measure 8 dimensions of health-related QOL. In addition, it includes a change self-assessment item that is not used in scoring. The instrument items cover: physical function, physical role, bodily pain, general health, vitality, social function, emotional role and mental health. The higher the score on the SF-36, the better the health.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University (Faculty of Physical Therapy), Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.